CLINICAL TRIAL: NCT05043480
Title: Pilot Study On Pulsed Electromagnetic Field Therapy For Osteosarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Louis Tee (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor-Investigator, Louis Tee, Senior Resident, Alexandra Hospital
Organization: Alexandra Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/01181
Record Dates: First submitted 2021-08-31; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Sarcopenia; Osteopenia or Osteoporosis
MeSH Terms: conditions — Sarcopenia; Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEMF arm (Experimental): In this single-arm study, all participants will be assigned to the intervention arm.
  Interventions: Device: PEMF

INTERVENTIONS:
Device: PEMF — Participants will receive pulsed electromagnetic fields (PEMF) exposure to alternate lower limbs weekly for 16 weeks. Participants will place alternate lower limb into the PEMF machine. Each lower limb will be exposed to 1.5mT magnetic field exposure for 10 mins once a week (total 10 min each week) for 16 weeks.

SUMMARY:
This prospective, single-site, single arm pilot study aims to assess the efficacy of Pulsed Electromagnetic Field (PEMF) exposure in the reduction of the decline in muscle strength, function and bone mineral density (BMD) in osteosarcopenia.

DETAILED DESCRIPTION:
This prospective, single-site, single-arm pilot study aims to assess the efficacy of Pulsed Electromagnetic Field (PEMF) exposure in the reduction of the decline in muscle strength, function and bone mineral density (BMD) in osteo-sarcopenia. For this pilot study, we will recruit 80 participants aged 65 years old and greater with osteo-sarcopenia, to receive PEMF therapy, at 1.5mT, once a week for 10 min to alternate lower limb (10 mins each week) weekly for 16 weeks. Participants will be followed up at baseline, 4, 8 and 12 and 17 weeks. At each follow-up, falls risk will be assessed by Short Physical Performance Battery (SPPB), including 6-minute walk and 5 sit-to-stand tests, Falls Efficacy Scale International (FESI), 3min-NS (3 minute Nutritional Screening) and SARC-F (Strength, Assistance with Walking, Rise from Chair, Climb Stairs and Falls) questionnaires. Muscle strength (hand grip and leg extension) and calf diameter are measured. Blood tests, saliva tests, and DEXA scans will be done at baseline, immediately after first PEMF exposure and week 17 to determine changes in biomarkers for senescence, bone/fat/muscle composition and skeletal muscle mass.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years old and above, which corresponds to the geriatric patient population seen at the Healthy Ageing clinics and wards
2. Diagnosed with primary osteopenia, including primary osteoporosis, by BMD measurements on DEXA scans
3. Diagnosed with sarcopenia by SARC-F
4. Willing and able to give written informed consent

Exclusion Criteria:

1. Presence of metallic implants, pacemakers or insulin pumps
2. Presence of rheumatological disease (such as osteoarthritis or rheumatoid arthritis)
3. Presence of secondary osteoporosis (such as hyperparathyroidism, steroid-induced osteoporosis)
4. Presence of end-stage organ failure, including severe dementia or cancer
5. Pregnant women

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower limb strength | 18 weeks
  Lower limb strength measurement measured by dynamometer
Handgrip strength | 18 weeks
  Handgrip strength measurement measured by dynamometer
Short Physical Performance Battery (SPPB) | 18 weeks
  Validated assessment tool for balance and lower limb strength (Score from 0 to 12)
6 minute walk test (6MWT) | 18 weeks
  Distance walked in a time of 6 minutes (units of meters)

SECONDARY OUTCOMES:
Lean muscle and fat mass | 18 weeks
  Lean muscle and fat mass measured by DEXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Santhosh Seetharaman, MBBS, Principal Investigator — Head of Department
Locations (1):
- Alexandra Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yap JLY, Tai YK, Frohlich J, Fong CHH, Yin JN, Foo ZL, Ramanan S, Beyer C, Toh SJ, Casarosa M, Bharathy N, Kala MP, Egli M, Taneja R, Lee CN, Franco-Obregon A. Ambient and supplemental magnetic fields promote myogenesis via a TRPC1-mitochondrial axis: evidence of a magnetic mitohormetic mechanism. FASEB J. 2019 Nov;33(11):12853-12872. doi: 10.1096/fj.201900057R. Epub 2019 Sep 13. PMID 31518158
- [Background] Parate D, Kadir ND, Celik C, Lee EH, Hui JHP, Franco-Obregon A, Yang Z. Pulsed electromagnetic fields potentiate the paracrine function of mesenchymal stem cells for cartilage regeneration. Stem Cell Res Ther. 2020 Feb 3;11(1):46. doi: 10.1186/s13287-020-1566-5. PMID 32014064
- [Background] Kurth F, Tai YK, Parate D, van Oostrum M, Schmid YRF, Toh SJ, Yap JLY, Wollscheid B, Othman A, Dittrich PS, Franco-Obregon A. Cell-Derived Vesicles as TRPC1 Channel Delivery Systems for the Recovery of Cellular Respiratory and Proliferative Capacities. Adv Biosyst. 2020 Nov;4(11):e2000146. doi: 10.1002/adbi.202000146. Epub 2020 Sep 2. PMID 32875708